CLINICAL TRIAL: NCT06036849
Title: Linking Physiological Responses to Clinical Outcomes Following Cervical Spine Manipulation: a Randomized Mechanistic Cross-over Trial
Brief Title: Linking Physiological Responses to Clinical Outcomes Following Cervical Spine Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Schweinhardt Petra, Prof. Dr. med., Balgrist University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CCRF Project
Record Dates: First submitted 2023-08-24; First posted 2023-09-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain
Keywords: Spinal Manipulation; Spinal Mobilization; Biomechanics; Physiological Responses; Clinical Outcomes
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: Randomized, mechanistic, cross-over clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to treatment allocation. It will not be possible to blind participants with respect to treatment allocation. However, participants will be blinded to the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neck pain participants: spinal manipulation first (Experimental): Spinal manipulation will be delivered first (followed by spinal mobilization at 72 hours).
  Interventions: Procedure: Spinal manipulation; Procedure: Spinal mobilization
- Neck pain participants: spinal mobilization first (Experimental): Spinal mobilization will be delivered first (followed by spinal manipulation at 72 hours).
  Interventions: Procedure: Spinal manipulation; Procedure: Spinal mobilization
- Healthy controls (No Intervention): Participants will attend a single session and no intervention will be performed but all experimental procedures will be identical to those occurring in the neck pain cohort. Measurements in individuals without neck pain are necessary for the assessment of potential baseline differences in the outcomes of interest between the patient cohort (with neck pain) and those without neck pain. Without this information, it is not possible to determine if the measured responses to spinal manipulation are due to the intervention or, systematic differences in the baseline outcomes of interest in the symptomatic cohort.

INTERVENTIONS:
Procedure: Spinal manipulation — The manipulation will be delivered to the articular pillar of the most painful level of the cervical spine, as determined by the patient history & physical examination, by a registered and practicing chiropractor. The participant will be positioned supine with the head supported by the clinician's hands. The articular process of the involved vertebra will be contacted by the antero-lateral aspect of the proximal phalanx of the second digit of the clinician's index finger. The head will be taken into flexion, ipsilateral lateral flexion and contralateral rotation to the pre-manipulative position. A rapid, controlled low-amplitude thrust will be applied in a further posterior-anterior line of drive. Ipsilateral in this instance means the same side as the primary contact i.e. for manipulation applied to the right side, the right side of the participant's neck will be contacted.
  Arms: Neck pain participants: spinal manipulation first; Neck pain participants: spinal mobilization first
Procedure: Spinal mobilization — The mobilization will consist of one set of posterior-anterior spinal mobilization applied with either a crossed-thumb or pisiform contact centrally over the spinous process of the most painful level of the cervical spine by a registered and practicing health care practitioner (i.e. physiotherapist).
  Arms: Neck pain participants: spinal manipulation first; Neck pain participants: spinal mobilization first

SUMMARY:
The investigators aim to investigate the relationship between delivery kinetics, physiological responses and clinical outcomes following spinal manipulation.

Neck pain participants will be randomised to attend two intervention sessions and will receive either a single cervical spine manipulation or mobilization (one set of central posterior-anterior mobilizations applied with either a crossed-thumb or pisiform contact) at the most painful level.

Participants without neck pain will attend a single experimental session, where all measurement procedures will be the same as for neck pain participants with the exception that no treatment will be delivered.

DETAILED DESCRIPTION:
For participants with neck pain, physiological responses & clinical outcomes associated with cervical spine manipulation and mobilization will be recorded. Both treatments will be delivered by several registered, practicing and experienced clinicians. A targeted history & physical examination will be conducted at the beginning of each experimental session to ensure it is ethical to proceed. Pre-treatment questionnaires regarding pain and treatment expectation will be completed. The participant will be instrumented with electromyographic and galvanic skin response sensors and required to wear a chest strap to measure heart rate variability. The participant will then lie in a quiet room for 10-15 minutes while baseline data is recorded. Following this, the treatment will be delivered & responses measured. After the treatment, the participant will again lie in a quiet room for 10-15 minutes while post-treatment data is recorded. Before leaving, all sensors will be removed and post-treatment questionnaires will be completed. The participant will return after 72 hours, at the same time of day, for the second session with the alternate treatment.

Participants without neck pain will attend a single experimental session, where all procedures will be the same as described above with the exception of treatment delivery and questionnaires describing neck pain changes following treatment.

Each visit will take approximately 2-3 hours and will be performed at the Balgrist University Hospital.

ELIGIBILITY:
Inclusion criteria:

All participants:

* 18-65 years of age
* English and/or French and/or German proficiency (to guarantee proper understanding of instructions and informed consent)
* Provision of informed consent

People with neck pain:

* Mechanical neck pain located inferior to the superior nuchal line and inferior border of the mandible and superior to the superior border of the clavicle, suprasternal notch and scapular spines bilaterally
* Neck pain of ≥ 12 weeks duration
* Neck pain not associated with an identified pathological cause
* Who have not received treatment for their neck pain (e.g. spinal manipulation, spinal mobilization, massage etc) in the previous 2 weeks

Exclusion criteria:

All participants:

* Unable to provide informed consent (e.g. due to language difficulties)
* Any neurological condition
* Any major medical or psychiatric condition (e.g. cardiovascular disease, diabetes, autoimmune disorders, major depressive disorder)
* Conditions and/or medications that could affect heart rate variability signals (e.g. hypertension, obesity (body mass index > 30), the current use of pain medications, steroids, antidepressants and/or β-blockers)
* Any chronic pain condition other than neck pain (e.g. low back pain)
* Pregnancy (all females will be asked verbally if there is a chance they are pregnant during screening)

People without neck pain:

* Acute pain
* Neck pain (> 3 consecutive days) in the last year

People with neck pain:

* Neck pain that does not originate from the cervical spine
* Who have received treatment for their neck pain (e.g. spinal manipulation, spinal mobilization, massage etc) in the previous 2 weeks
* Who have taken medication within the past 24 hours prior to the first visit and during their participation in the study
* All contraindications to the application of spinal manipulation and mobilization (e.g. personal or family history of a connective tissue disorder, current use of anticoagulant therapy, history of recent surgery and/or neck trauma, facial or intra-oral anesthesia or paresthesia, visual disturbances, dizziness and/or vertigo). Such contraindications will be screened during the medical history and physical examination performed by a registered health care clinician (e.g. chiropractor). Any participant not meeting the inclusion and exclusion criteria will be excluded from the study. As in routine daily clinical practice at the Balgrist University Hospital Chiropractic Polyclinic, the ultimate decision whether it is appropriate to deliver an intervention to the participant (spinal manipulation and/or mobilization) will be determined by the clinician delivering the treatment. The investigator is responsible for coordinating adequate medical care if complications occur. Possible subsequent medical care is contingent on the nature of the complication and could range from referral to the on-site Chiropractic Department Polyclinic for follow-up treatment of muscle soreness to referral to the Emergency Department of the Balgrist University Hospital (not expected).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Patient global impression of change following treatment | Immediately post intervention
  The self-report measure patient global impression of change reflects a patient's belief about the efficacy of treatment. It is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. It is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." Lower scores indicate better outcomes.
Change in numerical pain rating score | Immediately pre and immediately post intervention
  The numerical pain rating score is an 11-point pain scale, with 0 representing no pain and 10 representing the most intense pain tolerable. Participants are asked to rate their current pain on this scale. Larger change scores from pre to post-intervention indicate a greater reduction of pain.
Change in pressure pain threshold | Immediately pre and immediately post intervention
  Pressure pain thresholds are measured using an algometer (JTECH medical). The participant is instructed to say 'now' or 'stop' immediately when the sensation of pressure changes to pain. Lower values indicate a lower pain threshold and larger differences between pre and post-intervention measurements indicates greater changes in pain perception. Pressure pain thresholds will be performed bilaterally over the mastoid insertion of the sternocleidomastoid, the mid-belly of the upper trapezius and the upper third of the tibialis anterior three times, with the average used for statistical comparisons.
Change in active cervical spine range of motion | Immediately pre and immediately post intervention
  Active cervical spine range of motion is measured using a digital inclinometer (JTECH medical). The participant will be asked to move their head from a neutral position in a specified direction (i.e. flexion, extension, lateral flexion to both sides and rotation to both sides) as far as they are able. These movements will be performed (in each direction) three times, with the average used for statistical comparisons. Larger increases from pre to post-intervention indicate greater improvement in the participant's active range of motion.

SECONDARY OUTCOMES:
Electromyographic root-mean-squared magnitude | For 7 minutes pre-intervention, during the intervention (approximately 30 seconds) and for 7 minutes post-intervention
  Electromyographic root-mean-squared magnitudes are used to quantify the electrical activity of muscles. Bipolar sensors (Kendall) will be placed over specific portions of three muscles (sternocleidomastoid, upper trapezius and tibialis anterior) according to the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) guidelines. Larger root-mean-squared values indicate greater electrical activity of the muscle. Differences between pre and post-intervention resting values will be measured, allowing for a quantification of the electrical activity of the muscle. Additionally, the electrical activity of the muscle associated with spinal manipulation and mobilization will be measured during the intervention.
Change in heart rate variability | Immediately pre and immediately post intervention
  Heart rate variability measures the instantaneous change in heart rate. It is measured using a three-lead electrocardiogram protocol and a respiratory belt (ADInstruments). Larger variability in heart rate is reported to be associated with better health. Heart rate variability will be measured with the participant in 'quiet lying' pre and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Gorrell, PhD, Principal Investigator — University of Zürich and Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No